CLINICAL TRIAL: NCT05132426
Title: Osteopathic Manipulative Treatment for Recurrent Mastitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not receive sufficient funding and so no participants were recruited.
Sponsor: Western University of Health Sciences (Other)
Responsible Party: Principal Investigator, Brian Loveless, Chief Medical Officer, Western University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FB21/IRB/060
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Mastitis
Keywords: OMT; Mastitis
MeSH Terms: conditions — Mastitis | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial in which there will be a sham OMT control group and an OMT intervention group with a parallel group design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not be told whether they are enrolled in the OMT intervention group or the OMT Sham Group (placebo group). Investigators will be blinded to which participants are in each group and will collect data using only subject numbers provided on labels. Outcomes assessors will analyze data with coded patient data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMT Intervention Arm (Experimental): Myofascial release of the thoracic inlet is a treatment involving gentle pressure applied to shoulders and neck to move the tissue in different directions.
  Pectoral traction will have the doctor gently grasp and slowly pull the armpit area with a slow pulling force applied towards the shoulders.
  Diaphragm release with MFR consists of the doctor touching below the ribs on each side and gently applying pressure to move the tissue from side to side.
  Fascial release of the breast will have the doctor encircling the breast with their hands and inducing anterior traction. The doctor then induces motion in all directions. The doctor will then locate the affected spot and use a direct stripping motion from the base of the breast toward the areola until the restriction is released.
  Thoracic pump has the doctor placing their hands over the chest wall on each side and applying pressure and releasing pressure several times to generate a pumping action of about 100 times per minute.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)
- OMT Sham Arm (Sham Comparator): MFR of the thoracic inlet Sham: Operator's hands would encircle the thoracic inlet and would feel for somatic dysfunction in the area but would refrain from treating this area.
  Pectoral traction Sham: The doctor would contact the armpit area and diagnose the somatic dysfunction, but unlike the treatment group they would not do any treatment.
  Diaphragm release with MFR Sham: The doctor's hands are placed just below the ribcage and will feel for the direct restrictive barriers but will not augment the release.
  Fascial release of the breast Sham: The doctor would encircle the breast with their hands but would not induce motion or engage any direct barriers. The operator will find the barrier in the tissue but will refrain from treating it.
  Thoracic pump Sham: The doctor will hold their hands in place over the chest wall but will not try to affect the breathing motion and will not resist the upward motion of the rib cage during inhalation.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment (OMT) — Myofascial release of the thoracic inlet is a treatment involving gentle pressure applied to shoulders and neck to move the tissue in different directions.
  Pectoral traction will have the doctor gently grasp and slowly pull the armpit area with a slow pulling force applied towards the shoulders.
  Diaphragm release with MFR consists of the doctor touching below the ribs on each side and gently applying pressure to move the tissue from side to side.
  Fascial release of the breast will have the doctor encircling the breast with their hands and inducing anterior traction. The doctor then induces motion in all directions. The doctor will then locate the affected spot and use a direct stripping motion from the base of the breast toward the areola until the restriction is released.
  Thoracic pump has the doctor placing their hands over the chest wall on each side and applying pressure and releasing pressure several times to generate a pumping action of about 100 times per minute.

SUMMARY:
This study will investigate whether Osteopathic Manipulative Treatment (OMT) is effective in treating recurrent mastitis without the use of antibiotics and if it helps in preventing future recurrence of mastitis in individuals who have had multiple occurrences of mastitis.

DETAILED DESCRIPTION:
Lactational mastitis is a significant health issue for breastfeeding women, affecting up to 33% of this population. Mastitis is the most common reason cited for breastfeeding cessation among breastfeeding women. It is commonly treated with antibiotics, and some women will require multiple courses for recurrent episodes, which can lead to antibiotic resistance in the environment. The etiology of mastitis is incompletely defined in the literature, with sources describing an infectious or inflammatory condition. Osteopathic philosophy adds to this differential an examination of the musculoskeletal system, looking for a structure/function relationship. In this light, mastitis might be seen as a problem in the lymphatic system. An osteopathic physician would evaluate a patient for the presence of dysfunction in the fascial structures which drain the breast, and then apply osteopathic manipulative treatment (OMT) to address those dysfunctions. In patients with recurrent mastitis these dysfunctions in the fascia create an environment where impaired drainage leads to repeated episodes. The incorporation of OMT into those conservative treatments is proposed to improve the lymphatic drainage of the breast and therefore eliminate the need for antibiotic treatments. This study will investigate whether OMT is effective in treating recurrent mastitis without antibiotics, and in preventing future recurrence of mastitis in the same breast.

This will be a comparative effectiveness randomized pilot/feasibility clinical trial. We will be recruiting and treating participants who have had multiple diagnoses of mastitis in the same breast in the past 6 months. Participants must meet all inclusion/exclusion criteria in order to be enrolled in this study. Participants who are eligible for this study will undergo a standardized osteopathic examination that will be performed to evaluate connective tissue structures which drain the lymphatic system of the breast. The doctor will be looking for signs of somatic dysfunction which is described as changes in normal tissue qualities or body function that can be affected by osteopathic manipulation to improve health. Once somatic dysfunction is confirmed, patients will be randomly assigned to the sham-control group or the OMT intervention group. Both groups in the study will receive 24-48 hours of standard treatment for recurrent mastitis from their primary or referring physicians such as pain reduction, warm compresses, as well as management of overproduction of milk. If there are no improvements, then antibiotics may be given by their primary physician. If they are in the treatment group they will continue standard treatment but will also undergo OMT including myofascial release of the thoracic inlet, pectoral traction, diaphragm release with MFR, fascial release of the breast, and the thoracic lymphatic pump. If they are enrolled in the sham-control group they will receive sham treatments that will resemble the actual treatments but are not meant to be therapeutic. Both groups will be treated 3 times over 4 weeks, on week 1, week 2, and week 4. These treatments will be done by trained osteopathic physicians and medical students who are members of our osteopathic fellowship program.

Participants in both groups will be asked to take a global health assessment measured by the SF-36 (36-item Short Form Survey/RAND). This is a 36 question survey that will help to measure overall health outcomes during the entirety of the study. This will be taken at Day 0, the week 1 visit, the week 2 visit, the week 4 visit, and at the six-month follow up. In addition, after the initial visit, subjects will be asked to report if and when they have a recurrence of mastitis at any time during the course of the study, if and when they were unable to continue breastfeeding over the course of the study, and they will be asked to report if they experience any adverse effects from the treatment they receive. These data points will be taken at every visit and subjects will be asked to report any such instances to the research assistant if anything is experienced between research visits. The primary comparison will be standard treatment for recurrent mastitis patients with OMT sham versus standard treatment with the addition of OMT for recurrent mastitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 50 years old.
* Signed an informed consent form.
* Clinical diagnosis of recurrent mastitis: more than 2 episodes of lactational mastitis in the same breast in a 6-month time period.
* Evidence of somatic dysfunction upon undergoing an osteopathic structural exam.

Exclusion Criteria:

* Mammary abscesses.
* Health problems related to pregnancy.
* Inability to receive OMT due to open wounds, fractures, anuresis, necrotizing fasciitis, congestive heart failure, or unstable cardiac conditions.
* Less than 18 years of age or more than 50 years of age.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Mastitis in the sham-control group versus the OMT intervention group. | 6 months
  Comparing the number of individuals who have a recurrence of mastitis in the sham-control group versus the OMT intervention group.

SECONDARY OUTCOMES:
Global Health Assessment (SF-36 Survey) scores between the sham-control group and the OMT intervention group. | 6 months
  Comparing the results of 36-item Short Form Survey/RAND between the sham-control group and the OMT intervention group.
Continuation of breastfeeding between the sham-control group and the OMT intervention group. | 6 months
  Comparing the number of individuals who are able to continue breastfeeding in the sham-control group versus the OMT intervention group.
Evaluation of Safety based on adverse events between the sham-control group and the OMT intervention group. | 6 months
  Comparing and documenting the number of individuals who have adverse effects to OMT in sham-control group versus OMT intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Western University of Health Sciences, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No